CLINICAL TRIAL: NCT05439044
Title: A Real-World Study of Anti-SARS-CoV-2 Monoclonal Antibodies in Patients at High Risk of Severe Forms of Covid-19
Brief Title: A Real-World Study of Anti-SARS-CoV-2 Monoclonal Antibodies
Acronym: COVIMAB
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP220631
Record Dates: First submitted 2022-06-27; First posted 2022-06-30 (Actual); Last update posted 2022-07-08 (Actual); Status verified 2022-06

CONDITIONS: Immunocompromised Patients
Keywords: Covid-19; SARS-CoV-2; Immunocompromised; Monoclonal Antibodies; Mortality
MeSH Terms: conditions — COVID-19 | interventions — Data Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients who have received an anti-SARS-CoV-2 monoclonal antibody: Patients who have received an anti-SARS-CoV-2 monoclonal antibody, either prophylactically or curatively.
  Interventions: Other: Data collection

INTERVENTIONS:
Other: Data collection — Anti SARS-CoV-2 Monoclonal Antibodies: casirivimab-imdevimab (Ronapreve) OR bamlanivimab-etesevimab OR tixagevimab-cilgavimab (Evusheld) OR regdanvimab OR sotrovimab (Xevudy) OR adintrevimab

SUMMARY:
Absence of anti-SARS-CoV-2 vaccine response or insufficient vaccine response may occur in immunocompromised patients. Being at high risk of a severe form of Covid-19, they may be eligible to receive recombinant anti-SARS-CoV-2 monoclonal antibodies (mAbs). This study aims to describe patients who received anti-SARS-CoV-2 mAbs, in prophylaxis and/or curative of covid-19, and to analyze the hospitalization and mortality rates. This study is multicentric on all the university hospitals of Paris (AP-HP).

ELIGIBILITY:
Inclusion Criteria:

* Adult ≥ 18 years old
* Patients who received at least one administration of the following therapies: casirivimab-imdevimab, bamlanivimab-etesevimab, tixagevimab-cilgavimab, regdanvimab, sotrovimab or adintrevimab

Exclusion Criteria:

* Patients opposed to the collection of their personal data

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult hospital patients treated with anti-SARS-CoV-2 monoclonal antibodies.
Sampling Method: Non-Probability Sample
Enrollment: 4000 (Estimated)
Dates: Start 2020-03-01 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Mortality rate | 29 days after last administration
  Covid-19 mortality : Explore the mortality rate related to COVID-19 in patients treated with anti-SARS-CoV-2 monoclonal antibodies

SECONDARY OUTCOMES:
Hospitalizations rate | 29 days after last administration
  Explore the hospitalizations rate related to COVID-19 in patients treated with anti-SARS-CoV-2 monoclonal antibodies in prophylaxis
Mortality rate | 29 days after last administration
  Explore the mortality rate related to COVID-19 in patients treated with anti-SARS-CoV-2 monoclonal antibodies in prophylaxis
Hospitalizations rate | 90 days after last administration
  Explore the hospitalizations rate related to COVID-19 in patients treated with anti-SARS-CoV-2 monoclonal antibodies in prophylaxis
Mortality rate | 90 days after last administration
  Explore the mortality rate related to COVID-19 in patients treated with anti-SARS-CoV-2 monoclonal antibodies in prophylaxis
Hospitalizations rate | 29 days after last administration
  Explore the hospitalizations rate related to COVID-19 in patients treated with anti-SARS-CoV-2 monoclonal antibodies in healing
Mortality rate | 29 days after last administration
  Explore the mortality rate related to COVID-19 in patients treated with anti-SARS-CoV-2 monoclonal antibodies in healing
Hospitalizations rate | 90 days after last administration
  Explore the hospitalizations rate related to COVID-19 in patients treated with anti-SARS-CoV-2 monoclonal antibodies in healing
Mortality rate | 90 days after last administration
  Explore the mortality rate related to COVID-19 in patients treated with anti-SARS-CoV-2 monoclonal antibodies in healing
Proportion of hospitalizations | 29 days after last administration
  Proportion of hospitalizations from all causes, in patients treated prophylactically and curatively by anti-SARS-CoV-2 monoclonal antibodies
Proportion of deaths | 29 days after last administration
  Proportion of deaths from all causes, in patients treated prophylactically and curatively by anti-SARS-CoV-2 monoclonal antibodies
Proportion of hospitalizations | 90 days after last administration
  Proportion of hospitalizations from all causes, in patients treated prophylactically and curatively by anti-SARS-CoV-2 monoclonal antibodies
Proportion of deaths | 90 days after last administration
  Proportion of deaths from all causes, in patients treated prophylactically and curatively by anti-SARS-CoV-2 monoclonal antibodies

CONTACTS AND LOCATIONS:
Overall Officials: Jeremie Zerbit, PharmD, Principal Investigator — Pharmacy Department, Cochin Hospital, Assistance Publique des Hôpitaux de Paris (AP-HP)
Locations (1):
- Assistance Publique - Hôpitaux de Paris (AP-HP) - Cochin Hospital, Paris, Île-de-France Region, France

IPD SHARING:
Plan to Share IPD: No